CLINICAL TRIAL: NCT04641000
Title: The Alberta BLOOM Long Term Follow Up Study: The Microbiome of Preterm Children in Immune Development
Brief Title: The Alberta BLOOM Long Term Follow Up Study
Acronym: BLOOM-LTFU
Status: Terminated | Type: Observational
Why Stopped: The BLOOM-LTFU study has evolved into the ongoing BLOOM-PCS Study (REB20-1442).
Sponsor: University of Calgary (Other)
Collaborators: University of Alberta (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Marie-Claire Arrieta, Dr., University of Calgary
Other Study IDs: REB19-1780
Record Dates: First submitted 2020-11-17; First posted 2020-11-23 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Infant, Premature, Diseases; Infant; Asthma; Asthma in Children; Allergies; Infant, Extremely Premature
Keywords: Microbiota; Microbiome; Gastrointestinal Microbiome
MeSH Terms: conditions — Infant, Premature, Diseases; Asthma; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, observational clinical cohort study involving children born very preterm at less than 31 weeks and six days gestation. The purpose of this study is to investigate the microbiome (the collection of microbes in a biological site) alternations resulting from preterm birth and associations with the risk of immune dysregulation, asthma and allergies.

DETAILED DESCRIPTION:
One important factor in gut health is the large community of microbes (tiny living things such as bacteria) that live on the human body called the microbiome. Recent studies have shown that premature babies are more likely to have changes in their gut microbiome that are associated with health issues. However, the specific microbiome features that are involved in the development of premature babies is still unknown. Therefore, this study examines the impact of very premature birth on the baby's microbiome, and how microbiome alterations are involved in health issues such as immune dysregulation, allergies and asthma.

The large communities of microbes in the gut play a major role on the microbiome that will form during infancy and childhood. Factors such as diet, exposure to antibiotics, surgical procedures, and mode of delivery, can strongly affect the dynamics microbiome development. It is well known that microbiome alterations are associated with disorders such as asthma. However, the features involved in disease development and progression are highly understudied. Through this clinical study, we will evaluate associations between the early patterns of microbial colonization in premature infants and their risk to develop asthma later in childhood.

The hypothesis of the study is that microbial alterations resulting from preterm birth causally contribute to the allergy and asthma risk in infants (defined by atopic-wheeze) through immune mechanisms.

ELIGIBILITY:
Inclusion Criteria:

1. Born at ≤ 31 weeks + 6 days gestation (316/7 weeks);
2. Previously participated in the PROBIO and/or BLOOM PTN and/or BLOOM PTB research studies.
3. Provide a signed and dated informed consent form.
4. Willing and able to attend a clinic visit at Alberta Children's Hospital in Calgary, Alberta.
5. Parent/guardian providing consent must be able to speak and understand English.

Exclusion Criteria:

1. Has congenital gastrointestinal anomalies or has a history of gastrointestinal surgery.
2. Has major chromosomal anomalies.

Ages: 1 Year to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study recruits very early preterm infants that previously participated on at least one of the PROBIO, BLOOM PTN or BLOOM PTB studies.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2022-03-26 (Actual)

PRIMARY OUTCOMES:
Microbiome Establishment and Assembly | 1-2 Years Corrected Gestational Age
  Fecal microbial diversity and the relative abundance of bacterial and eukaryotic taxa, as assessed by polymerase chain reaction of the 16S and ITS2 gene and functional analysis on 16S taxonomic surveys for all participants from birth to around 1-year CGA. Changes in fecal microbial diversity and microbial population structures from birth to around 1-year CGA for all participants as assessed by shotgun metagenomics.
Metabolome | 1-2 Years Corrected Gestational Age
  Human and microbial metabolites as assessed by untargeted metabolomics, ultra-performance liquid chromatography ultrahigh-resolution Fourier transform (FT) combined with mass spectrometry to identify human and microbial metabolites for all participants from birth to around 1-year CGA.
Asthma Risk | 1-2 Years Corrected Gestational Age
  Health outcomes such as asthma risk that are influenced by novel linkages between gut microbiome features (taxonomical and functional) as assessed by the Asthma Predictive Index, which involves determining history of wheeze, atopic dermatitis, familial history and eosinophilia.
Allergies | 1-2 Years Corrected Gestational Age
  Skin reactivity to common allergens as assessed by a skin prick test.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Claire Arrieta, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada